CLINICAL TRIAL: NCT00767533
Title: Immunobiology of Cancer
Status: Terminated | Type: Observational
Why Stopped: PI left
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: VAR0033; SU-10012008-1313 (Other: Stanford University alternate IRB Number)
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To learn whether or not an Interferon defect in cell signaling, recently discovered in immune cells from melanoma patients as well as breast cancer patients, is common to all cancers.

DETAILED DESCRIPTION:
BACKGROUND

We have previously demonstrated that tumor-specific T cells could be identified in >50% of patients with metastatic melanoma and these cells appeared to be rendered anergic in vivo [Nature Medicine 5:677, 1999]. Recently we discovered that there is a signaling defect in the Interferon (IFN) pathway in immune cells from melanoma patients [PLOS Medicine 4:897 2007]. Interestingly, preliminary studies are showing the same defect in immune cells from breast cancer patients (unpublished). We would like to expand our research to all types of cancer to determine whether these phenomena occur in different cancer types.

OBJECTIVES

Our primary objective is to determine whether there is an IFN signaling defect in different types of cancers and to determine what is causing this defect.

The second objective is to determine whether these PBMCs are rendered anergic.

INVESTIGATIONAL PLAN

The study population will consist of patients who have been diagnosed with cancer, regardless of sex or ethnicity. Blood will be collected during the subjects regularly scheduled laboratory appointment and peripheral blood mononuclear cells (PBMCs) will be isolated for research purposes. These PBMCs will undergo studies, i.e. phosflow, qPCR, proliferation, survival, etc., to determine immune responses for T cells (CD4 and CD8), B cells (CD19), natural killer cells (CD16), and possibly monocytes (CD14).

ELIGIBILITY:
Inclusion Criteria:Participants who have cancer or participants who do not have cancer and/or an autoimmune disorder and are age 18 or over. Exclusion Criteria:Participants who have an autoimmune disorder and/or are under the age of 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have cancer or participants who do not have cancer and/or an autoimmune disorder and are age 18 or over.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2008-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter P Lee, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States